CLINICAL TRIAL: NCT06946394
Title: Application of Pegmolesatide in Renal Anemia: the Effectiveness and Safety of Switching to Two Different Regimens of Pegmolesatide in Patients With Non Dialysis CKD Treated With rhuEPO or HIF-PHI
Brief Title: Two Different Regiments of Pegmolesatide for Anemia in Patients With Chronic Kidney Disease Not Receiving Dialysis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSM-20039-402
Record Dates: First submitted 2024-11-10; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-07

CONDITIONS: Renal Anemia in Non-dialysis Chronic Kidney Disease
Keywords: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pegmolesatide optimize medication regimen group (Experimental): initial phase：Body weight ≤60kg, initial dose 2.0mg; Body weight > 60kg, initial dose 3.2mg, once every 4 weeks by subcutaneous injection.
  Adjustment phase：based on Hb levels and its changes every 4 weeks, once a month by subcutaneous injection.
  Interventions: Drug: Pegmolesatide
- Pegmolesatide standard medication regimen group (Active Comparator): initial phase：0.04mg/kg body weight, once every 4 weeks by subcutaneous injection.
  Adjustment phase：based on Hb levels and its changes every 4 weeks, once a month by subcutaneous injection.
  Interventions: Drug: Pegmolesatide

INTERVENTIONS:
Drug: Pegmolesatide — Pegmolesatide Injection: Specification 1mL: 4.0mg (National Medical Products Administration Approval No. H20230020), administered once every 4 weeks
  Other Names: EPO-018B

SUMMARY:
This was a multicenter, randomized, open label, non inferiority clinical study. It consisted of a 24-week treatment period (0-24 weeks) and a 24-week extension period (25-48 weeks). About 160 patients which had received Recombinant human erythropoietin (rHuEPO) or Hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI) treatment were randomized in a 1:1 ratio to receive Pegmolesatide with different administration regimens.

DETAILED DESCRIPTION:
This was a multicenter, randomized, open label, non inferiority clinical study. It consisted of a 24-week treatment period (0-24 weeks) and a 24-week extension period (25-48 weeks). About 160 patients were randomized in a 1:1 ratio to Pegmolesatide optimize medication regimen group and Pegmolesatide standard medication regimen group. Patients in the investigational group received 2.0 mg (in patients weighing ≤60 kg) or 3.2 mg (in patients weighing >60 kg) as the initial dose, the initial dose of the control group was 0.04mg/kg, then were adjusted for every 4 weeks based on Hb levels and its changes. The primary endpoint was the change in Hb levels from baseline in week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old, gender not limited;
2. Weight ≥ 45kg; Body Mass Index (BMI) ≥ 18.5kg/m^2;
3. Diagnosed with CKD ≥ 6 months and estimated glomerular filtration rate (eGFR) ≥ 15mL/min/1.73m^2 before enrollment, and<60 mL/min/1.73m^2 (estimated GFR using CKD-EPI formula), with no expected renal replacement therapy plan during the study period;
4. rHuEPO or HIF-PHI should be used for ≥ 4 weeks and ≤ 12 weeks;
5. During the 28days and 3days before randomization, with Hb ≥ 70g/L and < 110g/L;
6. Understand the research procedure and voluntarily sign an informed consent form (ICF) in writing.

Exclusion Criteria:

1. Known to have hematological disorders or other diseases that cause anemia other than chronic kidney disease (CKD), such as primary pure red cell aplasia (PRCA), homozygous sickle cell disease, thalassemia/Cooley's anemia, multiple myeloma, hemolytic anemia, and myelodysplastic syndrome, or malignant tumors;
2. Known to be allergic to iron agents or polyethylene glycol;
3. Received red blood cell or whole blood transfusion therapy within the three months prior to randomization;
4. Have received oral or intravenous immunosuppressive or glucocorticoid therapy within the 12 weeks prior to randomization;
5. Individuals with poor blood pressure control;
6. C-reactive protein ≥ 30mg/L within the first 3 days of randomization;
7. Pregnant and lactating women, women of childbearing age who have a positive urine β - HCG test result before the trial, or those who have a pregnancy plan during the study period;
8. Assessment of cardiac function level III or IV within the first 3 days of randomization;
9. Within the first 3 days of randomization, the liver function was assessed as Grade C;
10. Researchers believe that subjects with any other factors that are not suitable for participating in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes of mean Hb levels from baseline in the standard medication regimen group and the optimized medication regimen group at week 24 of the treatment period. | the 24th week of treatment.
  Baseline Hb was defined as the assessments of Hb during 3days prior to first dose of the study treatment. Mean Hb levels at week 24 of the treatment period (Hb at week 24) was defined as the mean of Hb at day 168±5 of the treatment period. Changes of mean Hb levels from baseline in the standard medication regimen group and the optimized medication regimen group at week 24 of the treatment period was calculated by subtracting the baseline Hb from Hb at week 24.

SECONDARY OUTCOMES:
Median time for two groups of Hb values to reach the target for the first time | during the 48 weeks of treatment.
  Median time for two groups of Hb values to reach the target for the first time.
Proportion of subjects with Hb levels meeting the standard in two groups at each follow-up point | during the 48 weeks of treatment.
  Proportion of subjects with Hb levels meeting the standard in two groups at each follow-up point.
Change of Hb from baseline at each follow-up point | during the 48 weeks of treatment.
  Change of Hb from baseline at each follow-up point.
Change of red blood cell count from baseline at each follow-up point | during the 48 weeks of treatment.
  Change of red blood cell count from baseline at each follow-up point.
Change of hematocrit from baseline at each follow-up point | during the 48 weeks of treatment.
  Change of hematocrit from baseline at each follow-up point.
the fluctuation of Hb values between the two groups after 24 weeks (Hb variability) | after the 24 weeks of treatment.
  It was defined as the coefficient of variation of Hb values after 24 weeks, which was calculated by dividing the SD (standard deviation) by the mean of Hb after the 24 weeks of treatment.
The types and average doses of anti-anemia drugs of the subjects reaching the Hb target at each follow-up time point | during the 48 weeks of treatment.
  The types and average doses of anti-anemia drugs of the subjects reaching the Hb target at each follow-up time point.
Cumulative number of dose adjustments for both groups of subjects in weeks 24 and 48 | the 24th and 48th week of treatment.
  Cumulative number of dose adjustments for both groups of subjects in weeks 24 and 48.
Therapeutic response of populations with different baseline characteristics to pegmolesatide | at the week 24 of treatment.
  Changes of mean Hb levels of populations with different baseline characteristics from baseline at week 24 of the treatment period.
Patient reported outcomes (PROs) at baseline and at week 24 in both groups | baseline and the 24th week of treatment
  Health Survey Scale at baseline and at week 24 in both groups.
All-cause death | during the 24/48 weeks of treatment.
  Number of all-cause death events during the 24/48 weeks of treatment.
Cardiovascular death | during the 24/48 weeks of treatment.
  Number of cardiovascular death events during the 24/48 weeks of treatment.
Cerebral infarction and myocardial infarction | during the 24/48 weeks of treatment.
  Number of Cerebral infarction and myocardial infarction events during the 24/48 weeks of treatment.
Receive regular renal replacement therapy | during the 24/48 weeks of treatment.
  Number of subjects receive regular renal replacement therapy during the 24/48 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Lin, M.D., Principal Investigator — The First Affiliated Hospital of Dalian Medical University

IPD SHARING:
Plan to Share IPD: No
The Principal Investigator have not yet considered when and in what form to share the data

REFERENCES:
- [Background] Zhang P, Jiang Y, Xu C, Zhou L, Zheng H, Xie D, Guo M, Huang X, Lu G, Jiang H, Qiu H, Liu B, Li S, Chen Q, Xia Y, Sun B, Yang X, Zhang S, Du S, Sun M, Chen M, Zhong A, Wang X, Zhao Z, Zhou H, Li G, Ren Y, Luo Q, Yang A, Luo P, Tang S, Xu C, Wang Q, Wang X, Yan T, He W, Qin S, Zhang W, Lv L, Wang C, Liu H, Li J, Wu Q, Pan C, Li C, He L, Chen J. Pegmolesatide for the treatment of anemia in patients undergoing dialysis: a randomized clinical trial. EClinicalMedicine. 2023 Oct 28;65:102273. doi: 10.1016/j.eclinm.2023.102273. eCollection 2023 Nov. PMID 37954906